CLINICAL TRIAL: NCT03892967
Title: Enhanced, EHR-Facilitated Cancer Symptom Control (E2C2) Trial
Brief Title: Enhanced, EHR-facilitated Cancer Symptom Control Pragmatic Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-007779; NCI-2020-06973 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015083 (NIH); UM1CA233033 (NIH); E2C2 (Other: Mayo Clinic Physical Medicine and Rehabilitation)
Record Dates: First submitted 2019-03-19; First posted 2019-03-27 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (interview) (Experimental): Patients randomized to E2C2 intervention participate in an interview over 30-45 minutes. Providers and stakeholders also participate in an interview over 15-30 minutes.
  Interventions: Other: Interview; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Interview — Participate in interview
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial investigates enhanced, electronic health record (EHR)-facilitated cancer system control. Cancer and its treatment are often associated with severe, disabling symptoms that have been causally linked to diminished survival, increased healthcare utilization, degraded quality of life, unemployment, and non-adherence to recommended cancer treatments. Collaborative case management for control of moderate or worse sleep disturbance, pain, anxiety, depression, fatigue (SPADE symptoms), and physical dysfunction among cancer survivors and patients with cancer may improve quality of life, symptom severity, and adherence to cancer treatment, and may also reduce need for acute care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a cluster randomized pragmatic trial with a stepped wedge design to test the hypothesis that a symptom control-focused enhanced, electronic health record (EHR)-facilitated cancer symptom control (E2C2) intervention will significantly reduce sleep disturbance, pain, anxiety, depression, fatigue (SPADE) symptom and physical dysfunction scores, reduce unplanned hospitalizations and emergency department visits, improve adherence to cancer therapies, and improve self-reported quality of life.

II. Evaluate the hypothesis that use of a multifaceted, evidence-based implementation strategy to support adoption and use of the E2C2 system will result in improvements in implementation and clinical outcomes.

III. Conduct a mixed methods evaluation to detect, understand and reduce disparities in the adoption and implementation of the E2C2 intervention among elderly and rural-dwelling patients with cancer.

OUTLINE:

The first Primary Objective involves a stepped wedge enrollment into the study intervention. Involvement is based off the patients' responses to the pain questionnaire (low pain = no involvement, moderate pain = offer of patient education materials, severe pain = involvement of a Symptom Care Manager). Symptom Care Managers will work with interested patients who endorse high pain to help address and manage their pain. The third objective involves a subset of patients included in the E2C2 who are offered to participate in a one-time interview lasting 30-45 minutes. Providers and stakeholders also will be invited to participate in an interview lasting 15-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Being seen for a solid or liquid cancer at a Midwest Mayo Clinic Midwest Mayo Clinic Health Systems (MCHS) site or for a solid tumor at Mayo Clinic Rochester

Exclusion Criteria:

* No Minors (under age 18) will receive the questionnaires but no further exclusions can be made based on the standard of care for questionnaire assignment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50207 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Cheville, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Finney Rutten LJ, Ruddy KJ, Chlan LL, Griffin JM, Herrin J, Leppin AL, Pachman DR, Ridgeway JL, Rahman PA, Storlie CB, Wilson PM, Cheville AL. Pragmatic cluster randomized trial to evaluate effectiveness and implementation of enhanced EHR-facilitated cancer symptom control (E2C2). Trials. 2020 Jun 5;21(1):480. doi: 10.1186/s13063-020-04335-w. PMID 32503661
- [Derived] Cheville AL, Herrin J, Pachman DR, Grzegorczyk V, Kroenke K, Ridgeway JL, Minteer SA, Austin JD, Griffin JM, Chlan L, Tofthagen C, Mitchell SA, Smith A, Ruddy KJ. Electronic health record-facilitated symptom surveillance and collaborative care intervention in oncology (E2C2): a cluster-randomised, population-level, stepped-wedge, pragmatic trial. Lancet Oncol. 2026 Jan;27(1):125-136. doi: 10.1016/S1470-2045(25)00526-1. Epub 2025 Dec 1. PMID 41344348
- [Derived] Minteer SA, Ridgeway JL, Pachman DR, Austin JD, Griffin JM, Ruddy KJ, Cheville AL. Barriers and facilitators to using practice facilitators to implement a remote cancer symptom management intervention: a mixed methods study. BMC Health Serv Res. 2025 Sep 3;25(1):1189. doi: 10.1186/s12913-025-13378-1. PMID 40903741
- [Derived] Kuharic M, Merle JL, Cella D, Mitchell SA, DiMartino L, Ridgeway JL, Dizon DS, Paudel R, Austin JD, Wong SL, Flores AM, Cheville AL, Smith JD; IMPACT Consortium. Psychometric evaluation of the NoMAD instrument in cancer care settings: assessing factorial validity, measurement invariance, and differential item functioning. Implement Sci Commun. 2025 Jun 16;6(1):72. doi: 10.1186/s43058-025-00756-3. PMID 40524282
- [Derived] Austin JD, Finney Rutten LJ, Fischer K, Ridgeway J, Minteer S, Griffin JM, Pachman DR, Ruddy KJ, Cheville A. Advancing Care Team Adoption of Electronic Health Record Systems for Cancer Symptom Management: Findings From a Hybrid Type II, Cluster-Randomized, Stepped-Wedge Trial. JCO Oncol Pract. 2025 Feb;21(2):209-217. doi: 10.1200/OP.24.00280. Epub 2024 Aug 6. PMID 39106420
- [Derived] Ridgeway JL, Cheville AL, Fischer KJ, Tesch NK, Austin JD, Minteer SA, Pachman DR, Chlan LL, Ruddy KJ, Griffin JM. Tracking activities and adaptations in a multi-site stepped wedge pragmatic trial of a cancer symptom management intervention. Contemp Clin Trials Commun. 2024 Feb 9;38:101269. doi: 10.1016/j.conctc.2024.101269. eCollection 2024 Apr. PMID 38380342
- [Derived] Kroenke K, Lam V, Ruddy KJ, Pachman DR, Herrin J, Rahman PA, Griffin JM, Cheville AL. Prevalence, Severity, and Co-Occurrence of SPPADE Symptoms in 31,866 Patients With Cancer. J Pain Symptom Manage. 2023 May;65(5):367-377. doi: 10.1016/j.jpainsymman.2023.01.020. Epub 2023 Feb 2. PMID 36738867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2019 to January 2023, 50,207 patients (in fifteen clusters) were enrolled and administered ePROMs in association with oncology visits.
Pre-assignment Details: Participants could be enrolled for more than one Period over the course of the study.
Units Other Than Participants: Clusters (provider groups)
Groups:
- Sequence 1: Sequence 1 began usual care on 4/1/2019 and entered EHR-facilitated collaborative care starting on 10/1/2019 (Step 2) until end of study on 1/31/2023
- Sequence 2: Sequence 2 began usual care on 4/1/2019 and entered EHR-facilitated collaborative care starting on 6/1/2020 (Step 3) until end of study on 1/31/2023
- Sequence 3: Sequence 3 began usual care on 4/1/2019 and entered EHR-facilitated collaborative care starting on 2/1/2021 (Step 4) until end of study on 1/31/2023
- Sequence 4: Sequence 4 began usual care on 4/1/2019 and entered EHR-facilitated collaborative care starting on 10/1/2021 (Step 5) until end of study on 1/31/2023
- Sequence 5: Sequence 5 began usual care on 4/1/2019 and entered EHR-facilitated collaborative care starting on 6/1/2022 (Step 6) until end of study on 1/31/2023
Period: Step 1: 4/1/2019-9/30/2019
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 2709; 3 Clusters (provider groups) | 4023; 3 Clusters (provider groups) | 4353; 3 Clusters (provider groups) | 3724; 3 Clusters (provider groups) | 1906; 3 Clusters (provider groups)
Answered >=1 Electronic Patient Reported Outcome Measure | 1992; 3 Clusters (provider groups) | 3098; 3 Clusters (provider groups) | 3314; 3 Clusters (provider groups) | 2967; 3 Clusters (provider groups) | 1467; 3 Clusters (provider groups)
Answered >=2 Electronic Patient Reported Outcome Measures (Analytic cohort: this subgroup was exposed to the full intervention and the effect of exposure could be assessed) | 1426; 3 Clusters (provider groups) | 2295; 3 Clusters (provider groups) | 2530; 3 Clusters (provider groups) | 2281; 3 Clusters (provider groups) | 1178; 3 Clusters (provider groups)
Completed (Trial participants who responded to at least two electronic patients reported outcome measures (ePROMs) were included in the primary analysis. We list those patients here as "completed." However, participants who completed one or more ePROMs were also included in secondary analyses evaluating individual symptom scores. Additionally, the entire trial cohort (N=50,207) were included in secondary utilization and survival analyses.) | 1426; 3 Clusters (provider groups) | 2295; 3 Clusters (provider groups) | 2530; 3 Clusters (provider groups) | 2281; 3 Clusters (provider groups) | 1178; 3 Clusters (provider groups)
Not Completed | 1283; 0 Clusters (provider groups) | 1728; 0 Clusters (provider groups) | 1823; 0 Clusters (provider groups) | 1443; 0 Clusters (provider groups) | 728; 0 Clusters (provider groups)
Not completed — Participants did not answer at least two surveys and were not included in the analytic cohort | 1283 | 1728 | 1823 | 1443 | 728
Period: Step 2: 10/1/2019-5/31/2020
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 1877; 3 Clusters (provider groups) | 2846; 3 Clusters (provider groups) | 3490; 3 Clusters (provider groups) | 2696; 3 Clusters (provider groups) | 1599; 3 Clusters (provider groups)
Answered >=1 Electronic Patient Reported Outcome Measure | 1615; 3 Clusters (provider groups) | 2420; 3 Clusters (provider groups) | 3121; 3 Clusters (provider groups) | 2382; 3 Clusters (provider groups) | 1445; 3 Clusters (provider groups)
Answered >=2 Electronic Patient Reported Outcome Measures (Analytic cohort: this subgroup was exposed to the full intervention and the effect of exposure could be assessed) | 1403; 3 Clusters (provider groups) | 2120; 3 Clusters (provider groups) | 2716; 3 Clusters (provider groups) | 2144; 3 Clusters (provider groups) | 1233; 3 Clusters (provider groups)
Completed (Trial participants who responded to at least two electronic patients reported outcome measures (ePROMs) were included in the primary analysis. We list those patients here as "completed." However, participants who completed one or more ePROMs were also included in secondary analyses evaluating individual symptom scores. Additionally, the entire trial cohort (N=50,207) were included in secondary utilization and survival analyses.) | 1403; 3 Clusters (provider groups) | 2120; 3 Clusters (provider groups) | 2716; 3 Clusters (provider groups) | 2144; 3 Clusters (provider groups) | 1233; 3 Clusters (provider groups)
Not Completed | 474; 0 Clusters (provider groups) | 726; 0 Clusters (provider groups) | 774; 0 Clusters (provider groups) | 552; 0 Clusters (provider groups) | 366; 0 Clusters (provider groups)
Not completed — Participants did not answer at least two surveys and were not included in the analytic cohort | 474 | 726 | 774 | 552 | 366
Period: Step 3: 6/1/2020-1/31/2021
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 2360; 3 Clusters (provider groups) | 3566; 3 Clusters (provider groups) | 4516; 3 Clusters (provider groups) | 3552; 3 Clusters (provider groups) | 1541; 3 Clusters (provider groups)
Answered >=1 Electronic Patient Reported Outcome Measure | 2047; 3 Clusters (provider groups) | 3058; 3 Clusters (provider groups) | 4121; 3 Clusters (provider groups) | 3221; 3 Clusters (provider groups) | 1413; 3 Clusters (provider groups)
Answered >=2 Electronic Patient Reported Outcome Measures (Analytic cohort: this subgroup was exposed to the full intervention and the effect of exposure could be assessed) | 1650; 3 Clusters (provider groups) | 2573; 3 Clusters (provider groups) | 3606; 3 Clusters (provider groups) | 2813; 3 Clusters (provider groups) | 1261; 3 Clusters (provider groups)
Completed (Trial participants who responded to at least two electronic patients reported outcome measures (ePROMs) were included in the primary analysis. We list those patients here as "completed." However, participants who completed one or more ePROMs were also included in secondary analyses evaluating individual symptom scores. Additionally, the entire trial cohort (N=50,207) were included in secondary utilization and survival analyses.) | 1650; 3 Clusters (provider groups) | 2573; 3 Clusters (provider groups) | 3606; 3 Clusters (provider groups) | 2813; 3 Clusters (provider groups) | 1261; 3 Clusters (provider groups)
Not Completed | 710; 0 Clusters (provider groups) | 993; 0 Clusters (provider groups) | 910; 0 Clusters (provider groups) | 739; 0 Clusters (provider groups) | 280; 0 Clusters (provider groups)
Not completed — Participants did not answer at least two surveys and were not included in the analytic cohort | 710 | 993 | 910 | 739 | 280
Period: Step 4: 2/1/2021-9/30/2021
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 1954; 3 Clusters (provider groups) | 3468; 3 Clusters (provider groups) | 4626; 3 Clusters (provider groups) | 3606; 3 Clusters (provider groups) | 1472; 3 Clusters (provider groups)
Answered >=1 Electronic Patient Reported Outcome Measure | 1660; 3 Clusters (provider groups) | 3028; 3 Clusters (provider groups) | 4259; 3 Clusters (provider groups) | 3273; 3 Clusters (provider groups) | 1328; 3 Clusters (provider groups)
Answered >=2 Electronic Patient Reported Outcome Measures (Analytic cohort: this subgroup was exposed to the full intervention and the effect of exposure could be assessed) | 1369; 3 Clusters (provider groups) | 2575; 3 Clusters (provider groups) | 3664; 3 Clusters (provider groups) | 2776; 3 Clusters (provider groups) | 1157; 3 Clusters (provider groups)
Completed (Trial participants who responded to at least two electronic patients reported outcome measures (ePROMs) were included in the primary analysis. We list those patients here as "completed." However, participants who completed one or more ePROMs were also included in secondary analyses evaluating individual symptom scores. Additionally, the entire trial cohort (N=50,207) were included in secondary utilization and survival analyses.) | 1369; 3 Clusters (provider groups) | 2575; 3 Clusters (provider groups) | 3664; 3 Clusters (provider groups) | 2776; 3 Clusters (provider groups) | 1157; 3 Clusters (provider groups)
Not Completed | 585; 0 Clusters (provider groups) | 893; 0 Clusters (provider groups) | 962; 0 Clusters (provider groups) | 830; 0 Clusters (provider groups) | 315; 0 Clusters (provider groups)
Not completed — Participants did not answer at least two surveys and were not included in the analytic cohort | 585 | 893 | 962 | 830 | 315
Period: Step 5: 10/1/2021-5/31/2022
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 1859; 3 Clusters (provider groups) | 3185; 3 Clusters (provider groups) | 4504; 3 Clusters (provider groups) | 3796; 3 Clusters (provider groups) | 1303; 3 Clusters (provider groups)
Answered >=1 Electronic Patient Reported Outcome Measure | 1639; 3 Clusters (provider groups) | 2796; 3 Clusters (provider groups) | 4119; 3 Clusters (provider groups) | 3495; 3 Clusters (provider groups) | 1161; 3 Clusters (provider groups)
Answered >=2 Electronic Patient Reported Outcome Measures (Analytic cohort: this subgroup was exposed to the full intervention and the effect of exposure could be assessed) | 1351; 3 Clusters (provider groups) | 2340; 3 Clusters (provider groups) | 3479; 3 Clusters (provider groups) | 3045; 3 Clusters (provider groups) | 1001; 3 Clusters (provider groups)
Completed (Trial participants who responded to at least two electronic patients reported outcome measures (ePROMs) were included in the primary analysis. We list those patients here as "completed." However, participants who completed one or more ePROMs were also included in secondary analyses evaluating individual symptom scores. Additionally, the entire trial cohort (N=50,207) were included in secondary utilization and survival analyses.) | 1351; 3 Clusters (provider groups) | 2340; 3 Clusters (provider groups) | 3479; 3 Clusters (provider groups) | 3045; 3 Clusters (provider groups) | 1001; 3 Clusters (provider groups)
Not Completed | 508; 0 Clusters (provider groups) | 845; 0 Clusters (provider groups) | 1025; 0 Clusters (provider groups) | 751; 0 Clusters (provider groups) | 302; 0 Clusters (provider groups)
Not completed — Participants did not answer at least two surveys and were not included in the analytic cohort | 508 | 845 | 1025 | 751 | 302
Period: Step 6: 6/1/2022-1/31/2023
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 2206; 3 Clusters (provider groups) | 3208; 3 Clusters (provider groups) | 4668; 3 Clusters (provider groups) | 3804; 3 Clusters (provider groups) | 1541; 3 Clusters (provider groups)
Answered >=1 Electronic Patient Reported Outcome Measure | 1940; 3 Clusters (provider groups) | 2828; 3 Clusters (provider groups) | 4233; 3 Clusters (provider groups) | 3487; 3 Clusters (provider groups) | 1329; 3 Clusters (provider groups)
Answered >=2 Electronic Patient Reported Outcome Measures (Analytic cohort: this subgroup was exposed to the full intervention and the effect of exposure could be assessed) | 1409; 3 Clusters (provider groups) | 2031; 3 Clusters (provider groups) | 3270; 3 Clusters (provider groups) | 2735; 3 Clusters (provider groups) | 1055; 3 Clusters (provider groups)
Completed (Trial participants who responded to at least two electronic patients reported outcome measures (ePROMs) were included in the primary analysis. We list those patients here as "completed." However, participants who completed one or more ePROMs were also included in secondary analyses evaluating individual symptom scores. Additionally, the entire trial cohort (N=50,207) were included in secondary utilization and survival analyses.) | 1409; 3 Clusters (provider groups) | 2031; 3 Clusters (provider groups) | 3270; 3 Clusters (provider groups) | 2735; 3 Clusters (provider groups) | 1055; 3 Clusters (provider groups)
Not Completed | 797; 0 Clusters (provider groups) | 1177; 0 Clusters (provider groups) | 1398; 0 Clusters (provider groups) | 1069; 0 Clusters (provider groups) | 486; 0 Clusters (provider groups)
Not completed — Participants did not answer at least two surveys and were not included in the analytic cohort | 797 | 1177 | 1398 | 1069 | 486

BASELINE CHARACTERISTICS:
Population: The accurate number of baseline participants in the analytic cohort is 24874. This is because 10390 participants contributed to both Usual Care and EHR-facilitated Collaborative Care. The numbers in the usual care (control) and EHR-facilitated collaborative care (intervention) columns accurately reflect the participants who contributed data to the comparator conditions. Unfortunately, we cannot make this distinction in the "total" column which is automatically calculated.
Groups:
- Usual Care (Control): Participants were administered ePROM surveillance alone.
- EHR-facilitated Collaborative Care (Intervention): Participants were administered ePROMs during EHR-facilitated collaborative care (ECC) periods. Automated responses, matched to symptom type and intensity, appeared following a patient's report of an actionable symptom, defined as >=4/10 on a numeric rating scale (NRS). For any actionable symptom, respondents were asked if they wanted to receive symptom-specific self-management resources. For severe symptoms, >=7/10, respondents were asked if they wanted to work remotely with a Symptom Care Manager (SCM) to develop an individualized symptom management plan.
- Total: Total of all reporting groups
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention) | Total
Number analyzed (Participants) | 16180 | 19084 | 35264
Age, Customized [Count of Participants; unit: Participants]
  Age: <=35 | 566 | 646 | 1212
  Age: 35-45 | 1200 | 1514 | 2714
  Age: 45-55 | 2336 | 2877 | 5213
  Age: 55-65 | 4188 | 4993 | 9181
  Age: 65-75 | 4933 | 5871 | 10804
  Age: 75-85 | 2466 | 2689 | 5155
  Age: >85 | 491 | 494 | 985
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9621 | 11138 | 20759
  Male | 6559 | 7946 | 14505
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15982 | 18816 | 34798
  Not Hispanic or Latino | 134 | 189 | 323
  Unknown or Not Reported | 64 | 79 | 143
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 62 | 86 | 148
  Asian | 248 | 357 | 605
  Native Hawaiian or Other Pacific Islander | 7 | 6 | 13
  Black or African American | 149 | 180 | 329
  White | 15468 | 18189 | 33657
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 246 | 266 | 512
Region of Enrollment [Number; unit: participants]
  United States | 16180 | 19084 | 35264

OUTCOME MEASURES:

1. Primary Outcome: Sleep Disturbance, Pain, Anxiety, Depression, Fatigue (SPADE) Symptom Scores.
Description: Measured by 11-point Numeric Rating Scales (NRS) for sleep disturbance, pain, anxiety, depression, fatigue, and physical function impairment at clinic encounters. Symptoms were assessed on a scale of 0 to 10 with higher scores indicating worse outcomes.
  Changes in sleep disturbance, pain, anxiety, depression, fatigue, and physical function impairment from baseline score were modeled jointly as a co-primary outcome.
Time Frame: Up to 46 months (beginning from a participants' index medical oncology encounter until death, last clinical encounter, or end of study)
Population: The analytic cohort includes trial participants who completed 2 or more NRS assessments.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention)
Number analyzed (Participants) | 16180 | 19084
score on a scale
  Anxiety | 2.09 [2.05 to 2.13] | 1.98 [1.94 to 2.02]
  Depression | 1.90 [1.86 to 1.93] | 1.81 [1.78 to 1.85]
  Fatigue | 3.27 [3.22 to 3.32] | 3.21 [3.15 to 3.26]
  Pain | 2.18 [2.12 to 2.24] | 2.14 [2.09 to 2.20]
  Impaired Physical Function | 2.75 [2.69 to 2.80] | 2.78 [2.72 to 2.84]
  Sleep | 2.46 [2.41 to 2.51] | 2.39 [2.34 to 2.44]

2. Primary Outcome: Physical Function Numerical Rating Scale (NRS) Scores
Description: Measured by 11-point Numeric Rating Scales (NRS) for sleep disturbance, pain, anxiety, depression, fatigue, and physical function impairment at clinic encounters. Symptoms were assessed on a scale of 0 to 10 with higher scores indicating worse outcomes.
  Changes in sleep disturbance, pain, anxiety, depression, fatigue, and physical function impairment following any NRS score of >=4/10 modeled jointly as a co-primary outcome.
Time Frame: as for outcome 1
Population: The analytic cohort includes trial participants who completed 2 or more NRS assessments and reported at least 1 NRS score >= 4/10
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention)
Number analyzed (Participants) | 9839 | 13084
units on a scale
  Anxiety | 2.51 [2.05 to 2.63] | 2.37 [2.24 to 2.49]
  Depression | 2.27 [2.14 to 2.40] | 2.17 [2.04 to 2.30]
  Fatigue | 3.96 [3.80 to 4.12] | 3.87 [3.72 to 4.03]
  Pain | 2.53 [2.37 to 2.69] | 2.55 [2.39 to 2.70]
  Physical function impairment | 3.23 [3.05 to 3.42] | 3.30 [3.11 to 3.48]
  Sleep | 2.91 [2.75 to 3.06] | 2.85 [2.70 to 3.01]

3. Secondary Outcome: Change in Anxiety Score
Description: Measured PROMIS-CAT T-scores up to every four months, depending on visit frequency. A T-score of 50 represents the average score for the U.S. general population, with a standard deviation of 10. A higher score indicates a worse outcome. PROMIS-CAT T-scores were averaged for the control and intervention periods.
Time Frame: Baseline to 46 months
Population: Patients who answered >=1 Anxiety PROMIS-CAT were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention)
Number analyzed (Participants) | 19952 | 25970
score on a scale | 51.86451 (9.036415) | 51.35445 (9.303022)

4. Secondary Outcome: Change in Depression Score
Description: Measured PROMIS-CAT T-score up to every four months, depending on visit frequency. A T-score of 50 represents the average score for the U.S. general population, with a standard deviation of 10. A higher score indicates a worse outcome. PROMIS-CAT T-scores were averaged for the control and intervention periods.
Time Frame: Baseline to 46 months
Population: Patients who answered >=1 Depression PROMIS-CAT were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention)
Number analyzed (Participants) | 19979 | 25498
score on a scale | 49.05267 (8.642265) | 48.49032 (8.666607)

5. Secondary Outcome: Change in Average Pain Interference Over the Past Week
Description: as for outcome 4
Time Frame: Baseline to 46 months
Population: Patients who answered >=1 Pain Interference PROMIS-CAT were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention)
Number analyzed (Participants) | 20225 | 26516
score on a scale | 52.57027 (9.80923) | 53.2717 (9.918807)

6. Secondary Outcome: Change in Physical Function Score
Description: Measured PROMIS-CAT up to every four months, depending on visit frequency. A T-score of 50 represents the average score for the U.S. general population, with a standard deviation of 10. A higher score indicates a better outcome. PROMIS-CAT T-scores were averaged for the control and intervention periods.
Time Frame: Baseline to 46 months
Population: Patients who answered >=1 Physical Function PROMIS-CAT were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention)
Number analyzed (Participants) | 20070 | 26239
score on a scale | 43.83007 (9.641792) | 43.18325 (9.561469)

7. Secondary Outcome: Health Care Utilization
Description: ER visits, hospitalizations, and ICU admissions
Time Frame: Up to 46 months (beginning from a participants' index medical oncology encounter until death, 18 months after last clinical encounter, or end of study)
Population: Utilization data were available for the entire E2C2 trial cohort irrespective of ePROM completion. To assess robustness, we conducted analyses that included the full cohort, the >=1 ePROM completers, and the >=2 ePROM completers. In addition, we created subgroups based on residential proximity to a trial site to assess the extent of care provided at non-participating institutions. Here we report the patients who completed 1 or more surveys and resided within 120 miles from a trial site.
Measure: Number; unit: events
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention)
Number analyzed (Participants) | 13090 | 15220
events
  Hospitalizations | 3415 | 3009
  ED visits | 4331 | 3495
  ICU admissions | 940 | 722

8. Secondary Outcome: Adherence to Cancer Treatment
Description: Number of doses of docetaxel and cyclophosphamide administered.
Time Frame: Up to 46 months (beginning from a participants' index medical oncology encounter until death or end of study)
Population: The analyses were restricted to the subgroup of patients with breast cancer being treated with docetaxel/cyclophosphamide in order to ensure comparable receipt of chemotherapeutic regimens between the comparator groups. Because docetaxel and cyclophosphamide may be first-/second-line therapy for breast cancer, a large participant subgroup that offered adequate power was chosen. Patients who crossed over from usual care to EHR-facilitated collaborative care were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: number of doses administered
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention)
Number analyzed (Participants) | 198 | 128
number of doses administered
  Number of doses of docetaxel administered | 3.530303 (1.088281) | 3.765625 (0.6458148)
  Number of doses of cyclophosphamide administered | 3.707071 (0.973151) | 3.78125 (0.7310601)

9. Secondary Outcome: Number of Deceased Participants
Description: Vital status (living or deceased) was determined by Accurint record search across multiple sources, including the Social Security Death Index
Time Frame: Up to 46 months (beginning from a participants' index medical oncology encounter until death or end of study)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention)
Number analyzed (Participants) | 16180 | 24874
Participants | 2214 | 3192

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for up to 46 months (beginning from a participants' index medical oncology encounter until death or end of study) for all participants
Groups:
- Usual Care (Control): Participants were administered ePROM surveillance alone. Participants who responded to >=2 ePROMs were included in the analytic cohort.
- EHR-facilitated Collaborative Care (Intervention): Participants were administered ePROMs during EHR-facilitated collaborative care (ECC) periods. Automated responses, matched to symptom type and intensity, appeared following a patient's report of an actionable symptom, defined as >=4/10 on a numeric rating scale (NRS). For any actionable symptom, respondents were asked if they wanted to receive symptom-specific self-management resources. For severe symptoms, >=7/10, respondents were asked if they wanted to work remotely with a Symptom Care Manager (SCM) to develop an individualized symptom management plan.
  Participants who responded to >=2 ePROMs were included in the analytic cohort.
Arm/Group | Usual Care (Control) | EHR-facilitated Collaborative Care (Intervention)
All-Cause Mortality (participants affected / at risk) | 2214/16180 | 3192/24874
Serious Adverse Events (participants affected / at risk) | 0/16180 | 0/24874
Other Adverse Events (participants affected / at risk) | 0/16180 | 0/24874

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT03892967/Prot_SAP_020.pdf